CLINICAL TRIAL: NCT05692518
Title: Creation of Side-to-Side Compression Anastomosis Using the GT Metabolic Solutions DI Bio-fragmentable Magnetic Anastomosis System to Achieve Duodeno-Ileostomy Diversion in Adults With Obesity and Type 2 Diabetes Mellitus
Brief Title: MagDI Diversion Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: GTM-005
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, single-arm, feasibility device study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MAGNET System, DI Bio-fragmentable (Experimental): GT Metabolic Solutions DI Bio-fragmentable Magnetic Anastomosis System
  Interventions: Device: MAGNET System, DI Bio-fragmentable

INTERVENTIONS:
Device: MAGNET System, DI Bio-fragmentable — Anastomoses achieved by magnetic compression.

SUMMARY:
The purpose of this clinical research study is to evaluate the feasibility of the GT Metabolic Solutions DI Bio-fragmentable Magnetic Anastomosis System (MAGNET System, DI Bio-fragmentable) for creation of a side-by-side anastomosis duodeno-ileostomy in obese adults.

DETAILED DESCRIPTION:
The purpose of this clinical research study is to evaluate the feasibility of the GT Metabolic Solutions DI Bio-fragmentable Magnetic Anastomosis System (MAGNET System, DI Bio-fragmentable) for creation of a side-to-side anastomosis duodeno-ileostomy in obese adults. This partial diversion of intestinal contents from duodenum to the ileum is intended to facilitate weight management/loss in obese adults with type 2 diabetes mellitus (T2DM) and improve metabolic outcomes in obese adults with type 2 diabetes mellitus (T2DM). Side-by-side anastomoses are currently created by sutures, staples, and anastomotic compression devices. A predicate procedure is the single-anastomosis duodeno-ileostomy (SADI) procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age, inclusive, at the time of informed consent
2. BMI 30-35 kg/m2
3. Type 2 diabetes mellitus (T2DM), defined as HbA1c > 6.5%, without previous sleeve gastrectomy, and without plan to perform a concurrent sleeve gastrectomy.
4. Agrees to refrain from any type of additional bariatric or reconstructive surgery that would affect body weight for the duration of the study
5. If a child-bearing female, subject must commit to not becoming pregnant and agree to use contraception for the duration of the study
6. Willing and able to comply with protocol requirements

Exclusion Criteria:

1. Type 1 diabetes
2. Use of injectable insulin
3. Uncontrolled T2DM
4. Previous sleeve gastrectomy procedure or plan to perform a sleeve gastrectomy with the duodeno-ileal anastomosis procedure
5. Uncontrolled hypertension, dyslipidemia or sleep apnea
6. Prior intestinal, colonic or duodenal surgery, other than bariatric
7. Prior surgery, trauma, prostheses, disease or genetic expression which prevent or contra-indicate the procedure, including scarring and abnormal anatomy.
8. Refractory gastro-esophageal reflux disease (GERD)
9. Barrett's disease
10. Helicobacter pylori positive and/or active ulcer disease
11. Large hiatal hernia
12. Inflammatory bowel or colonic diverticulitis disease
13. Any anomaly precluding orogastric access by gastroscope and catheters, and manipulation techniques.
14. Implantable pacemaker or defibrillator
15. Psychiatric disorder, except well-controlled depression with medication for > 6 mo
16. History of substance abuse
17. Woman who is either pregnant or breast feeding
18. Woman of childbearing potential who does not agree to use an effective method of contraception.
19. Any comorbidity or current status of subject's physiological fitness that in the surgeon's or anesthesiologist's opinion represents safety concerns that make the subject medically unfit for the procedure.
20. Any anomaly preventing/contraindicating laparoscopic access and general laparoscopic procedures
21. Had surgical or interventional procedure within 30 days prior to procedure
22. Any scheduled surgical or interventional procedure planned within 30 days post-procedure
23. Any stroke/transient ischemic attack (TIA) within 6 months prior to consent
24. Requires chronic anticoagulation therapy (except aspirin)
25. Active infections requiring antibiotic therapy, unless resolved before undergoing the study procedure
26. Unable to comply with the follow-up schedule and assessments
27. Recent tobacco or nicotine product cessation within < 3 months prior to informed consent
28. Known allergies to the device components or contrast media
29. Limited life expectancy due to terminal disease
30. Currently participating in another clinical research study with an investigational drug or medical device
31. A positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2 or COVID-19) test prior to the study procedure in accordance with local COVID-19 protocol
32. Any condition that, in the investigator's opinion, may preclude completion of follow-up assessments through Day 360 (e.g., a medical condition that may increase the risk associated with study participation or may interfere with interpretation of study results, inability to adhere to the visit schedule, or poor compliance with treatment regimen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Creation of a patent anastomosis | 30 Days
  Confirmed radiologically or fluoroscopically

CONTACTS AND LOCATIONS:
Locations (1):
- Innova Medical Center, Tbilisi, Georgia, Georgia